CLINICAL TRIAL: NCT00924261
Title: Age-Related Gait Changes and Hip Flexibility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: D. Casey Kerrigan, M.D., M.S., University of Virginia, Department of Physical Medicine and Rehabilitation
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 10101; 5R01AG27192-3; 5R01AG027192 (NIH)
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Gait; Flexibility
Keywords: hip; gait; walking; falls; stretching; Flexibility; Aged

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hip Stretching (Experimental): Kneeling Hip flexor stretch - 3 minutes a day, daily, for 10 weeks
  Interventions: Other: Hip Stretch
- Shoulder Stretch (Experimental): Shoulder Stretch - 3 minutes daily for 10 weeks
  Interventions: Other: Shoulder Stretch

INTERVENTIONS:
Other: Hip Stretch — Hip flexor stretch daily for 3 min x 10 weeks
  Other Names: Thomas Test; Hip flexibility
  Arms: Hip Stretching
Other: Shoulder Stretch — Shoulder Adduction stretch - 3 minutes, daily, for 10 weeks
  Other Names: Shoulder Horizontal Adduction Stretch
  Arms: Shoulder Stretch

SUMMARY:
Based on their preliminary quantitative gait findings suggesting that limited passive hip extension range is a key functionally limiting impairment affecting gait, the investigators propose a supervised, specific stretching exercise with the aim to improve both peak hip extension and overall gait performance. While one goal is to demonstrate that reduced peak passive hip extension is a key, functionally significant, but reversible, impairment another is to improve our understanding of the relationship between impairment, functional limitation and gait ability.

DETAILED DESCRIPTION:
1. Test the hypothesis that both passive and dynamic hip extension during comfortable and fast walking speeds are reduced in the elderly groups compared to passive and dynamic peak hip extension in healthy young adults.
2. Test the hypothesis, separately for each elderly group, controlling for co-factors, that there is greater change in step length in the treatment group compared to the control group, after controlling for co-variates. We also expect greater changes in dynamic hip peak extension, a reduction in anterior pelvic tilt, improvement in age-related reductions in peak ankle plantar flexion and ankle power generation, and in dynamic CoM-CoP moment arm during both comfortable and fast walking, and an increase in comfortable walking speed.
3. Test the hypothesis separately for the frail elderly group who cannot independently perform IADL only, controlling for co-factors, that there is a greater change in secondary, non quantitative gait-parameters of the Timed Get Up and Go Test, Activities of Daily Living, Instrumental ADL function, fear of falling and number of falls during 6 months following intervention.
4. Test the hypothesis that the created forward dynamic model can accurately predict in individual subjects, the actual effect of an increase in passive peak hip extension on dynamic peak hip extension, anterior pelvic tilt, peak ankle plantar flexion and step length.

ELIGIBILITY:
Inclusion Criteria:

Healthy Elderly Adult Subjects:

1. 100 subjects aged 65 years and older will be recruited from the Charlottesville area.
2. Participants will be asked to fill out a health questionnaire identical to that used for all preliminary studies. This questionnaire verifies that the participants meet the inclusion criteria for the proposed research project.
3. After this initial health questionnaire screening, each participant will undergo a face-to-face history and physical examination screening.

Frail Elderly Subjects:

1. 100 subjects aged 65 years and older who meet the criteria of not being able to function independently, which is considered to be frail, living within the greater Charlottesville area will be recruited for participation in the study.

Exclusion Criteria:

Healthy Elderly:

1. acute medical illness,
2. diagnosis or symptoms of unstable angina or congestive heart failure,
3. pulmonary diagnosis or symptoms of emphysema, chronic obstructive disease or asthma and shortness of breath as a result of pulmonary diagnosis brought about by walking on a flat surface,
4. advanced cancer,
5. neurologic diagnosis including Parkinson's Disease, stroke, brain injury, cerebellar disease, myelopathy, myopathy, peripheral neuropathy, or active radiculopathy,
6. major orthopedic diagnosis in the lower back, pelvis, or lower extremities, including hip or other fracture since the age of 50, fused joint, joint replacement, or amputation,
7. severe osteoarthritis or rheumatoid arthritis or active joint or musculoskeletal pain in the back or lower extremities occurring at rest or with walking,
8. severe osteoporosis with a history of a fragility fracture occurring in the past 12 months, and
9. regular use of an assistive device for walking.

Exclusion criteria per physical examination will be:

1. physical signs of congestive heart failure,
2. muscle weakness (less than 4/5 manual muscle test strength in lower extremities or focal findings of 1/5 strength difference between sides or upper and lower extremities), absent knee extensor reflexes or positive Babinski responses,
3. corrected visual acuity worse than 20/100 or presence of a field defect,
4. poor mental state defined with a Mini-Mental Status Examination score less than or equal to 24/30,133
5. orthostatic hypotension (greater than 20mmHg decline in systolic blood pressure from supine to standing at one minute), and
6. unilateral sensory deficit in lower extremities, bilateral sensory loss in stocking distribution, proprioception less than 75% correct in identifying great toe position, or vibration (from with a 128Hz tuning fork) perceived for less than 10 seconds at either the great toe or medial malleolus in either extremity.

Frail Elderly (who do not Function Independently):

1. are unable to walk independently (i.e., unable to walk without the assistance of another person), or
2. have either an acute medical condition or a chronic underlying medical condition which would make it unfeasible or unsafe to participate.
3. Regular use of an assistive device, such as a cane, for walking is not an exclusion criterion as long as:

   * when using the device, the subject does not require the assistance of another person and
   * the subject can walk without the assistive device (with supervisory, but not physical assistance if needed) for the length of the testing walkway, ten times (with rest periods between) at both his/her comfortable walking speed and at a faster walking speed.
4. Based upon the questionnaire or medical history, the following specific exclusion criteria will be used:

   * acute medical illness,
   * symptoms of angina or dyspnea brought about by walking on a flat surface,
   * hip or knee replacement surgery or hip fracture in the previous six months,
   * advanced cancer and/or life expectancy of less than 12 months,
   * dementia or other illness characterized by cognitive impairment.
5. Based upon physical examination, subjects will be excluded if they have:

   * physical signs of congestive heart failure,
   * cognitive impairment defined as a Mini-Mental Status Examination score less than or equal to 24/30133 or
   * orthostatic hypotension (greater than 20mm Hg decline in systolic blood pressure from supine to standing at one minute).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Hip Extension | 10 weeks

SECONDARY OUTCOMES:
Hip Flexibility | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diedre C Kerrigan, MD, MS, Principal Investigator — University of Virginia
Locations (1):
- Department of Physical Medicine and Rehabilitation, University of Virginia, Charlottesville, Virginia, United States